CLINICAL TRIAL: NCT05033054
Title: Effect of SGLT2i on Cardiovascular Biomarkers in Patients With Type 2 Diabetes and CKD Stage 3b-4
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Robert Toto, PROFESSOR, University of Texas Southwestern Medical Center
Other Study IDs: STU-2021-0492
Record Dates: First submitted 2021-08-26; First posted 2021-09-02 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Kidney Disease, Chronic; Diabetes
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum CPP, Magnesium, creatinine, Klotho, HsCRP, PTH, FSF23. Urine Klotho, creatinine, Ngal,8-isoprostane. 24 hour urine FEMg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 1: Group 1: take prescribed SGLT2i after baseline visit.
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — Participants will ingest a standard dose of SGLT2i prescribed by the standard of care physician.

SUMMARY:
This is a prospective, observational study to assess the effect of SGLT2 inhibitors on surrogate markers of kidney and cardiovascular health in patients with stage 3b and 4 chronic kidney disease (CKD).

This study includes three clinic in person visits and weekly telephone visits for 12 weeks.

1. Recruit 28 patients with CKD stages 3b-4 and follow up for 12 weeks
2. Determine the effect of interventions on the primary outcome variable serum klotho measured by immunoprecipitation-immunoblot

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* All races and ethnicities
* All genders
* Type 2 diabetes mellitus
* History of hypertension defined as > 130 or > 80 mmHg or normotensive on pharmacologic therapy
* Estimated glomerular filtration rate (GFR) (CKD Epi equation) of 15-44 ml/min/1.73 m2 (Stages 3b-4 CKD)
* Urinary albumin creatinine ratio of > 200 mg/g <5000mg/g
* Ability of study participant or legally authorized representative to provide informed written consent
* Able to maintain stable dose of any vitamin D and any calcium supplements for 180 days post randomization.

Exclusion Criteria:

* Autosomal dominant or autosomal recessive polycystic kidney disease, lupus nephritis or anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis
* Receiving cytotoxic therapy, immunosuppressive therapy or other immunotherapy for primary or secondary renal disease within 6 months prior to enrolment
* History of organ transplantation
* Receiving therapy with a sodium glucose co-transporter 2 (SGLT2) inhibitor within 8 weeks prior to enrolment or previous intolerance of an SGLT2 inhibitor
* Type 1 diabetes (T1D)
* Active use of SGLT2 inhibitor
* History of persistent hypercalcemia (serum total Calcium > 10.5 mg/dl)
* Body mass index > 45 kg/m2
* Active on kidney transplant list
* Inability to provide informed consent
* Any condition outside the renal and cardiovascular disease area, such as but not limited to malignancy, with a life expectancy of less than 2 years based on investigator´s clinical judgement
* Active malignancy requiring treatment at the time of screening (with the exception of successfully treated basal cell or treated squamous cell carcinoma).
* Hepatic impairment (aspartate transaminase [AST] or alanine transaminase [ALT] >3x the upper limit of normal [ULN]; or total bilirubin >2x ULN at time of enrolment)
* Women of child-bearing potential (ie, those who are not chemically or surgically sterilized or who are not post-menopausal) who are not willing to use a medically accepted method of contraception that is considered reliable in the judgment of the investigator or women who have a positive pregnancy test at enrolment or randomization or women who are breast-feeding
* Participation in another clinical study with an investigational product (IP) during the last month prior to Enrolment
* Inability of the patient, in the opinion of the investigator, to understand and/or comply with procedures and/or follow-up OR any conditions that, in the opinion of the investigator, may render the patient unable to complete the study. Patients who cannot complete the patient reported outcome (PRO) assessments can still participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with type 2 diabetes mellitus and stage 3b-4 chronic kidney disease.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Change in serum klotho levels at 6 weeks | Baseline, 6 weeks
  Change in serum klotho levels in participants with advanced Diabetic Kidney Disease (DKD) at 6 weeks are measured by immunoprecipitation-immunoblot.
Change in serum klotho levels at 12 week | Baseline, 12 weeks
  Change in Serum klotho levels in participants with advanced Diabetic Kidney Disease (DKD) at 12 weeks are measured by immunoprecipitation-immunoblot.

SECONDARY OUTCOMES:
Change in serum magnesium levels at 6 weeks | Baseline, 6 weeks
  Mean change from baseline in serum magnesium levels at 6 weeks is measured. Serum magnesium levels are measured by measuring the level of magnesium in the blood.
Change in serum magnesium levels at 12 weeks | Baseline, 12 weeks
  Mean change from baseline in serum magnesium levels at 12 weeks is measured. Serum magnesium levels are measured by measuring the level of magnesium in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Toto, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No